CLINICAL TRIAL: NCT03565536
Title: Prospective Study of Nexavar for Neoadjuvant Treatment of Anaplastic Thyroid Cancer
Brief Title: Nexavar for Neoadjuvant Treatment of Anaplastic Thyroid Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fujian Medical University (Other)
Responsible Party: Principal Investigator, Bo Wang,MD, clinical professor, Fujian Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UTC-NEXAVAR
Record Dates: First submitted 2018-05-26; First posted 2018-06-21 (Actual); Last update posted 2024-04-19 (Actual); Status verified 2024-04

CONDITIONS: Thyroid Cancer, Anaplastic
Keywords: Nexavar; Anaplastic Thyroid Cancer; Neoadjuvant Treatment
MeSH Terms: conditions — Thyroid Carcinoma, Anaplastic | interventions — Sorafenib; Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Nexavar neoadjuvant treatment group (Experimental): After the patient had diagnosed as anaplastic thyroid cancer, Nexavar was used for neoadjuvant treatment. At 1 month and 2 months after treatment, it was assessed whether surgery could be performed.
  operation for possible surgical treatment,with complete thyroidectomy and cervical lymph node dissection are performed to completely resect thyroid tissue and metastatic lymphatic tissue.
  then External radiation therapy after surgery.
  Interventions: Drug: Nexavar; Procedure: operation; Radiation: External radiation therapy

INTERVENTIONS:
Drug: Nexavar — for Unresectable tumors ,After the patient had diagnosed as anaplastic thyroid cancer, Nexavar 400mg Bid was used for neoadjuvant treatment. At 1 month and 2 months after treatment, it was assessed whether surgery could be performed.
  Other Names: Nexavar neoadjuvant treatment group
Procedure: operation — If computed tomography (CT) evaluates for possible surgical treatment, complete thyroidectomy and cervical lymph node dissection are performed to completely resect thyroid tissue and metastatic lymphatic tissue.
Radiation: External radiation therapy — As the successful surgery, then continue on the basis of taking on Nexavar plus external beam radiation therapy

SUMMARY:
Undifferentiated thyroid cancer is the most malignant tumor of the thyroid gland, with a median survival of only 3 months. Most undifferentiated cancers lose the chance of surgery when they are first diagnosed. The current study, Nexavar, is used only for dedifferentiated thyroid cancer and has not been applied to undifferentiated cancer. This study attempted to apply it to preoperative treatment of undifferentiated cancer to see if it would shrink the tumor and give the patient an opportunity for surgery.

DETAILED DESCRIPTION:
Undifferentiated thyroid cancer is the most malignant tumor of the thyroid gland, with a median survival of only 3 months. Most undifferentiated cancers lose the chance of surgery when they are first diagnosed. The current study, Nexavar, is used only for dedifferentiated thyroid cancer and has not been applied to undifferentiated cancer. This study attempted to apply it to preoperative treatment of undifferentiated cancer to see if it would shrink the tumor and give the patient an opportunity for surgery.

We chose patients with recurrent or inoperable anaplastic thyroid cancer and used NEXAVAR for 1 month of neoadjuvant therapy. If tumor lesions begin to resolve, they continue neoadjuvant therapy until the end of the second month. The total duration of preoperative treatment is two months.at the end of the second month, a CT scan was performed to assess whether surgery could be performed. If surgery is possible, NEXAVAR will continue to perform adjuvant radiotherapy after the surgery.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Undifferentiated or poorly differentiated thyroid cancer
* Tumor invades the trachea, esophagus or common carotid artery that are Unresectable.
* Locally recurrent anaplastic thyroid cancer
* The lesion size is greater than 3cm
* Patients in whom the oncologist has decide to start therapy with NEXAVAR.

Exclusion Criteria:

* Lesions cannot be evaluated by imaging
* Synonymous with contraindications to Nexavar.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2020-12-30 (Actual); Study Completion 2020-12-30 (Actual)

PRIMARY OUTCOMES:
Thyroglobulin | Change from Baseline Blood Thyroglobulin at 1 month, 2 months, 3 months after treatment with NEXAVAR
  Thyroglobulin
CT assessment | Change from Baseline Blood Thyroglobulin at 1 month, 2 months, 3 months after treatment with NEXAVAR
  Maximum tumor diameter measured by CT
Length of contact surface between tumor and common carotid artery | Change from Baseline Blood Thyroglobulin at 1 month, 2 months, 3 months after treatment with NEXAVAR
  Length of contact surface between tumor and common carotid artery
Percentage of patients in whom the actual dose of sorafenib equaled the planned dose | 6 months after treatment with NEXAVAR
  Percentage of patients in whom the actual dose of sorafenib equaled the planned dose
MST | 12 months after treatment with NEXAVAR
  Median Survival Time (MST) was defined as the duration from the date of patient recruited to the date of death from any cause

SECONDARY OUTCOMES:
Overall tolerability of treatment as measured by rate of adverse events | 3 months after treatment with NEXAVAR
  Overall tolerability of treatment as measured by rate of adverse events
ORR | 1 month, 2 months, 3 months after treatment with NEXAVAR
  Overall Response Rate (ORR) was defined as the total of CR (Complete Response) and PR (Partial Response). CR and PR were assessed by independent reviewers according to the Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1. ORR evaluated in 1 to 3 months after treatment with NEXAVAR
TTP | 12 months after treatment with NEXAVAR
  Time to Progression (TTP) was defined as the duration from the date of patient recruited to the first progress at any site or the date of death
Rate of III-IV grade adverse events | 12 months after treatment with NEXAVAR
  Adverse events was evaluated during received protocol therapy according to CTCAE 4.03

CONTACTS AND LOCATIONS:
Locations (1):
- Fujian Medical University Union Hospital, Fuzhou, Fujian, China

IPD SHARING:
Plan to Share IPD: No